CLINICAL TRIAL: NCT05665634
Title: Brain Stimulation and Electroencephalography Pilot Study
Brief Title: Concurrent TMS and EEG Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00233571
Record Dates: First submitted 2022-12-19; First posted 2022-12-27 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Healthy
MeSH Terms: interventions — Electroencephalography

STUDY DESIGN:
Intervention Model Description: Within-subject design. Each participant will undergo the same TMS/EEG procedures twice with one week in between sessions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All participants (Experimental)
  Interventions: Device: Concurrent transcranial magnetic stimulation and electroencephalogram

INTERVENTIONS:
Device: Concurrent transcranial magnetic stimulation and electroencephalogram — Single and paired-pulse TMS will be applied to 5 different brain regions during simultaneous recording of EEG. Paired-pulse stimulations will have either 3 ms or 11 ms between pulses, to stimulate cortical inhibition and excitation respectively. Stimulation intensity for single-pulse stimulation blocks will be 120% of the resting motor threshold (RMT). For paired-pulse blocks, the conditioning (first) pulse will be delivered at a stimulation intensity of 80% RMT, and the test (second) pulse will be delivered at 120% RMT. Each test block will consist of 60 TMS trials and will last for 5 minutes. Order of test blocks will be pseudo-randomized across participants. Out of 5 stimulation sites, 3 will be determined based on individual's own brain anatomy and resting state connectivity. These 3 regions will be stimulated using all 3 TMS protocols. The other two regions will be determined based on the literature and only be targeted using the single pulse TMS protocol.

SUMMARY:
This study will investigate the test-retest reliability of transcranial magnetic stimulation (TMS) -evoked potentials (TEPs) as measured by electroencephalography (EEG), using three different TMS protocols over five different brain regions in healthy volunteers. The goal is to compare the test-retest reliability of single pulse, inhibitory and excitatory TMS protocols as well as two distinct targeting approaches. The main questions to answer are:

1. This study will investigate whether the test-retest reliability of TEPs differ across TMS protocols.
2. This study will investigate whether the test-retest reliability of TEPs differ between individualized and non-individualized targeting approaches.

DETAILED DESCRIPTION:
Participants will first undergo functional magnetic resonance imaging (fMRI) scanning where structural and resting-state functional images will be obtained. In two separate sessions, participants will attend two concurrent TMS/EEG session with one week in between.

During the TMS/EEG sessions, an EEG cap will be placed on the participant's head and the resting motor threshold will be obtained to calibrate the TMS intensity required for the stimulation of target regions. Once setup procedures are complete, eleven total blocks of TMS with simultaneous EEG recording will take place. Among eleven blocks, five of will use single-pulse stimulation (to stimulate cortical excitation), three will use paired-pulse stimulation with 3ms between pulses (to stimulate cortical inhibition), and three will use paired-pulse stimulation with 11ms between pulses (to stimulate greater cortical excitation). Five different brain regions will be targeted: three individualized targets either derived anatomically (motor cortex) or based on the individual's resting-state functional connectivity (dorsolateral prefrontal cortex and angular gryus) and two regions that are based on the literature (dorsolateral prefrontal cortex and angular gryus).

ELIGIBILITY:
Inclusion Criteria:

* Medically and psychiatrically healthy
* Between the ages of 18 and 65 years old
* Fluent in English and capable of providing informed consent
* Willing to remove any jewelry, hair clips, bobby pins, or any other potentially conducting or magnetic objects worn on or near the head

Exclusion Criteria:

* Weight greater than 350 lbs (the weight limit of the specialized TMS/EEG chair)
* Current serious medical or psychiatric illness, or recent heart disease
* Acute intoxication with any drug of abuse, including alcohol or cannabis
* Pregnancy
* History of neurological problems, including epilepsy, seizures, syncope, tinnitus, migraine, or frequent non-migraine (e.g. tension) headaches
* History of head trauma associated with loss of consciousness
* Language or hearing impairment that would undermine communication regarding consent, study procedures, and overall volunteer safety.
* Irritable skin
* For those undergoing MRI procedures in the current study: Any standard MRI contraindication (including implanted medical devices, metal in the body, or claustrophobia incompatible with MRI procedures)
* TMS-contraindicated medical devices, including cochlear implants, pacemaker, neurosensory stimulator, implantable defibrillator, insulin pump, clips, stents, or shunts that may be disrupted by or interact with TMS coil operation
* Taking medications that lower seizure threshold (see Appendix A: List of Contraindicated Medications)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Comparison of interclass correlation coefficients (ICC) of TMS Evoked Potential amplitudes, as measured by EEG, between single and paired-pulse TMS protocols | Session 1 and session 2 with one week between sessions
  TMS evoked potentials (TEP) during single and paired-pulse protocols will be measured by simultaneous EEG recording. TEP amplitudes at approximately 40, 60, 100 and 200 ms will be calculated per subject, individualized brain region (anatomically based M1, connectivity based DLPFC and angular gyrus), TMS protocol and session. ICCs will be calculated across sessions and subjects per TEP for each individualized brain region and TMS protocol. ICCs per brain region will be compared between single and paired-pulse TMS protocols.
Comparison of interclass correlation coefficients (ICC) of TMS Evoked Potential amplitudes, as measured by EEG, between individualized and non-individualized targeting approaches | Session 1 and session 2 with one week between sessions
  TMS evoked potentials (TEP) during single pulse TMS protocols will be measured by simultaneous EEG recording. TEP amplitudes at approximately 40, 60, 100 and 200 ms will be calculated per subject, individualized and non-individualized (connectivity-based vs literature-based DLPFC and angular gyrus) brain region and session. ICCs will be calculated across sessions and subjects per TEP for all brain regions (connectivity-based vs literature-based DLPFC and angular gyrus) that were targeted by single-pulse protocols. ICCs will be compared between individualized and non-individualized targeting approaches.

CONTACTS AND LOCATIONS:
Overall Officials: Fred Barrett, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No